CLINICAL TRIAL: NCT05489549
Title: Identifying Subclinical Transthyretin Cardiac Amyloidosis in Asymptomatic Carriers of the V122I TTR Allele
Brief Title: Subclinical Transthyretin Cardiac Amyloidosis in V122I TTR Carriers
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: The Cleveland Clinic (Other); Columbia University (Other); The University of Texas at Arlington (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Justin Grodin, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU-2022-0404; 1R01HL160892-01A1 (NIH)
Record Dates: First submitted 2022-07-29; First posted 2022-08-05 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Amyloidosis, Hereditary; Amyloidosis Cardiac; Amyloidosis, Familial; Transthyretin-Related (ATTR) Familial Amyloid Cardiomyopathy; Transthyretin Gene Mutation
Keywords: Amyloidosis; Transthyretin Amyloidosis; V122I TTR; p.Val142Ile TTR; Cardiac magnetic resonance imaging
MeSH Terms: conditions — Amyloidosis, Familial; Amyloid Neuropathies, Familial; Amyloidosis; Amyloidosis, Hereditary, Transthyretin-Related

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Venous blood will be collected by phlebotomy at enrollment for all participants. Both plasma and serum will be isolated and aliquoted for storage. Peripheral blood mononuclear cells will also be aliquoted in CPT tubes for generation of human-induced pluripotent stem cells and blood will also be aliquoted into PAXgene blood RNA tubes for future studies. All samples will be immediately frozen and stored until use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- V122I TTR carriers: Carriers and controls will undergo standardized, detailed CMRI assessments to test the hypothesis that V122I TTR carrier status will be associated with greater evidence of pathological amyloid progression in comparison with non-carriers.
  In addition to the CMRI assessments, carriers and controls enrolled at UT Southwestern will undergo standardized exercise CMRI assessments during the same study visit.
  V122I TTR carriers will undergo detailed biomarker assessments. These will be compared with controls and patients with symptomatic V122I hATTR-CA .
- Age-, sex-, and race-matched non-carrier controls: Carriers and controls will undergo standardized, detailed CMRI assessments to test the hypothesis that V122I TTR carrier status will be associated with greater evidence of pathological amyloid progression in comparison with non-carriers.
  In addition to the CMRI assessments, carriers and controls enrolled at UT Southwestern will undergo standardized exercise CMRI assessments during the same study visit.
  Controls will undergo detailed biomarker assessments. These will be compared with V122I TTR carriers and patients with symptomatic V122I hATTR-CA .
- Patients with symptomatic V122I hATTR-CA: Patients with symptomatic V122I hATTR-CA will undergo detailed biomarker assessments. These will be compared with V122I TTR carriers and controls.

SUMMARY:
Approximately 1.5 million of the 44 million Blacks in the United States are carriers of the valine-to-isoleucine substitution at position 122 (V122I) in the transthyretin (TTR) protein. Virtually exclusive to Blacks, this is the most common cause of hereditary cardiac amyloidosis (hATTR-CA) worldwide. hATTR-CA leads to worsening heart failure (HF) and premature death. Fortunately, new therapies that stabilize TTR improve morbidity and mortality in hATTR-CA, especially when prescribed early in the disease. However, hATTR-CA is often diagnosed at an advanced stage and conventional diagnostic tools lack diagnostic specificity to detect early disease.

The overall objectives of this study are to determine the presence of subclinical hATTR-CA and to identify biomarkers that indicate amyloid progression in V122I TTR carriers. The central hypothesis of this proposal is that hATTR-CA has a long latency period that will be detected through subclinical amyloidosis imaging and biomarker phenotyping.

The central hypothesis will be tested by pursuing 2 specific aims: Aim 1) determine the association of V122I TTR carrier status with CMRI evidence of amyloid infiltration; Sub-aim 1) determine the association of V122I TTR carrier status with cardiac reserve; Aim 2) determine the association between amyloid-specific biomarkers and V122I TTR carrier status; and Sub-aim 2) determine the association of amyloid-specific biomarkers with imaging-based parameters and evaluate their diagnostic utility for identifying subclinical hATTR-CA. In Aim 1, CMRI will be used to compare metrics associated with cardiac amyloid infiltration between a cohort of V122I TTR carriers without HF formed by cascade genetic testing and age-, sex-, and race-matched non-carrier controls. For Sub-Aim 1, a sub-sample of carriers and non-carrier controls enrolled in Aim 1 will undergo novel exercise CMRI to measure and compare cardiac systolic and diastolic reserve. Aim 2 involves measuring and comparing amyloid-specific biomarkers in V122I TTR carriers without HF with samples matched non-carriers (both from Aim 1) and individuals with symptomatic V122I hATTR-CA from our clinical sites. These biomarkers detect and quantify different processes of TTR amyloidogenesis and include circulating TTR, retinol binding protein 4, TTR kinetic stability, and misfolded TTR oligomers. Sub-aim 2 will establish the role of these biomarkers to detect imaging evidence of subclinical hATTR-CA disease.

ELIGIBILITY:
(V122I TTR carriers (or matched non-carriers))

Inclusion Criteria:

* Men and women ages 30-80 who are V122I TTR carriers (or matched non-carriers) without history of HF (this will be assessed by study personnel) and defined as: a) No history of hospitalization within the previous 12 months for management of HF; b) Without an elevated B-type natriuretic peptide level ≥100 pg/mL or NT-proBNP ≥360 pg/mL within the previous 12 months; or c) No clinical diagnosis of HF from a treating clinician
* Signed informed consent

Exclusion Criteria:

* A self-reported history or clinical history of HF
* Other known causes of cardiomyopathy
* History of light-chain cardiac amyloidosis
* Prior type 1 myocardial infarction (non-ST segment elevation myocardial Infarction {NSTEMI} or ST-elevation myocardial infarction {STEMI})
* Cardiac transplantation
* Body weight >250 lbs
* Estimated glomerular filtration rate ≤30 mL/min/1.73 m2
* Inability to safely undergo CMRI

(For participants with symptomatic V122I hATTR-CA, we will enroll probands with HF from Aim 1 or patients with suspected symptomatic V122I hATTR-CA from the three study sites.)

Inclusion Criteria:

* Men and women ages 30-80 who have symptomatic V122I hATTR-CA as determined by a history of HF (this will be assessed by study personnel) and defined as: a) History of hospitalization within the previous 12 months for management of HF; b) An elevated B-type natriuretic peptide level ≥100 pg/mL or NT-proBNP ≥360 pg/mL within the previous 12 months; or c) A clinical diagnosis of HF from a treating clinician.
* Have an established or suspected diagnosis of hATTR-CA based on either a) Biopsy confirmed by Congo red (or equivalent) staining with tissue typing with immunohistochemistry or mass spectrometric analysis or immunoelectron microscopy, OR b) positive technetium-99m (99mTc)-pyrophosphate or -bisphosphonate scan, combined with accepted laboratory criteria without abnormal M-protein.
* TTR gene sequencing that is pending or that is confirming the V122I variant
* Signed informed consent

Exclusion Criteria:

* Other known causes of cardiomyopathy
* History of light-chain cardiac amyloidosis
* Cardiac transplantation
* Liver transplantation
* Previous treatment with a TTR stabilizer (tafamidis, acoramidis) within the prior 14 days or TTR any silencer (inotersen, patisiran, eplontersen)
* Estimated glomerular filtration rate ≤30 mL/min/1.73 m2

Ages: 30 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: For Aim 1, the will be a cross-sectional cohort study of 200 V122I TTR carriers and 200 age-, sex- and race-matched non-carrier controls without heart failure.
  For Sub-aim 1, this will be a cross-sectional sub-study of the 2 groups enrolled in Aim 1 at UT Southwestern.
  For Aim 2, this will be a cross-sectional cohort study of 200 V122I TTR carriers without HF (see Aim 1, Approach), 200 age-, sex-, and race-matched controls (see Aim 1), and 100 patients with symptomatic V122I hATTR-CA who will undergo detailed biomarker assessments.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
(Aim 1) Evidence of amyloid infiltration as measured by ECV | At baseline (for V122I TTR carriers and age-, sex-, and race-matched controls)
  ECV expansion represents interstitial expansion from amyloid infiltration and greater levels can distinguish amyloidosis from other hypertrophic cardiomyopathies and correlate with cardiac amyloidosis disease severity.
(Sub-aim 1) Δ stroke volume index (ΔSVi) | At baseline (for V122I TTR carriers and age-, sex-, and race-matched controls) enrolled at UT Southwestern
  We will measure and compare ΔSVi (%) from rest to peak stress in V122I TTR carriers and non-carrier controls. Participants will exercise within the bore of the magnet using an MR compatible ergometer with adjustable electronic resistance (Ergospect Cardio-Stepper, Ergospect). Cardiac imaging will be performed at rest and during exercise at 25% (low intensity), 50% (moderate intensity), and 66% (heavy intensity) of maximal predicted work rate. Workloads will be maintained for ~5 min at each stage - 3 min to achieve a physiological steady-state and then 2 minutes for image acquisition.

SECONDARY OUTCOMES:
(Aim 1) Late gadolinium enhancement | At baseline (for V122I TTR carriers and age-, sex-, and race-matched controls)
  We will use a PSIR sequence, limiting operator-dependency. Global subendocardial enhancement, transmural LGE, and focal, patchy LGE are all features of cardiac amyloidosis, representing interstitial expansion. In cardiac amyloidosis, unlike other cardiomyopathies, LGE is correlated to amyloid infiltration not interstitial fibrosis.
(Aim 1) Native T1 and T2 mapping | At baseline (for V122I TTR carriers and age-, sex-, and race-matched controls)
  Native T1 and T2 mapping represent diffuse interstitial expansion and myocardial edema, respectively. Native T1 measurements are abnormally elevated in amyloidosis and much higher in comparison with other cardiomyopathies that may be associated with interstitial expansion.
(Aim 1) Post-gadolinium T1 signal intensity | At baseline (for V122I TTR carriers and age-, sex-, and race-matched controls)
  Post-gadolinium T1 signal intensity changes characteristically with myocardial signal nulling before the blood pool signal in amyloidosis (opposite of non-amyloid hearts). We will test for this characteristic pattern using a Look-Locker "TI Scout" sequence.
(Aim 1) High resolution cardiac cine imaging for cardiac morphology | At baseline (for V122I TTR carriers and age-, sex-, and race-matched controls)
  High resolution cardiac cine imaging will measure cardiac morphology in all 4 chambers of the heart.
(Aim 1) High resolution cardiac cine imaging for global systolic function as ejection fraction | At baseline (for V122I TTR carriers and age-, sex-, and race-matched controls)
  High resolution cardiac cine imaging will measure cardiac systolic function in all 4 chambers of the heart by assessing ejection fraction.
(Aim 1) High resolution cardiac cine imaging for global systolic function as fractional area change | At baseline (for V122I TTR carriers and age-, sex-, and race-matched controls)
  High resolution cardiac cine imaging will measure cardiac systolic function in all 4 chambers of the heart by assessing fractional area change.
(Aim 1) High resolution cardiac cine imaging for global systolic function via novel feature tracking | At baseline (for V122I TTR carriers and age-, sex-, and race-matched controls)
  High resolution cardiac cine imaging will measure cardiac systolic function in all 4 chambers of the heart using novel feature tracking methods.
(Aim 1) High resolution cardiac cine imaging for global diastolic function via novel feature tracking. | At baseline (for V122I TTR carriers and age-, sex-, and race-matched controls)
  High resolution cardiac cine imaging will measure cardiac diastolic function in all 4 chambers of the heart using novel feature tracking methods.
(Aim 1) LV strain from magnetic resonance tissue tagging | At baseline (for V122I TTR carriers and age-, sex-, and race-matched controls)
  Magnetic resonance tissue tagging is the gold-standard for measuring LV strain and strain rate, providing highly sensitive measures of subclinical systolic and diastolic function.
(Aim 1) Phase contrast MRI to assess diastolic function by measurement of mitral inflow velocities. | At baseline (for V122I TTR carriers and age-, sex-, and race-matched controls)
  Phase contrast MRI will be used to assess LV diastolic function by assessing the ratio of early (E) and late (A) mitral inflow velocities which can be abnormal in V122I TTR carriers which can be abnormal in V122I TTR carriers.
(Aim 1) Phase contrast MRI to assess diastolic function by calculating the E/e' strain rate. | At baseline (for V122I TTR carriers and age-, sex-, and race-matched controls)
  Phase contrast MRI will be used to assess LV diastolic function by cine feature tracking and MR tissue tagging to calculate the E/e' strain rate which can be abnormal in V122I TTR carriers.
(Sub-aim 1) End diastolic volume index (EDVi, ml/m2) in all 4 chambers | At baseline (for V122I TTR carriers and age-, sex-, and race-matched controls) enrolled at UT Southwestern
  Exercise CMRI will be performed immediately following the resting CMRI protocol described for the Sub-aim 1 primary outcome.
(Sub-aim 1) End systolic volume index (ESVi, ml/m2) in all 4 chambers | At baseline (for V122I TTR carriers and age-, sex-, and race-matched controls) enrolled at UT Southwestern
  Exercise CMRI will be performed immediately following the resting CMRI protocol described for the Sub-aim 1 primary outcome.
(Sub-aim 1) Stroke volume index (SVi, ml/m2, ΔSVi is the primary outcome) in all 4 chambers | At baseline (for V122I TTR carriers and age-, sex-, and race-matched controls) enrolled at UT Southwestern
  Exercise CMRI will be performed immediately following the resting CMRI protocol described for the Sub-aim 1 primary outcome.
(Sub-aim 1) Ejection fraction (LVEF, %) in all 4 chambers | At baseline (for V122I TTR carriers and age-, sex-, and race-matched controls) enrolled at UT Southwestern
  Exercise CMRI will be performed immediately following the resting CMRI protocol described for the Sub-aim 1 primary outcome.
(Sub-aim 1) Longitudinal strain (LS, %) | At baseline (for V122I TTR carriers and age-, sex-, and race-matched controls) enrolled at UT Southwestern
  Exercise CMRI will be performed immediately following the resting CMRI protocol described for the Sub-aim 1 primary outcome.
(Aim 2) TTR concentration | At baseline for all three cohorts
  Venous blood will be collected by phlebotomy at enrollment for all participants. Both plasma and serum will be isolated and aliquoted for storage. Plasma TTR levels will be measured with commercially available ELISA assays.
(Aim 2) RBP4 concentration | At baseline for all three cohorts
  Venous blood will be collected by phlebotomy at enrollment for all participants. Both plasma and serum will be isolated and aliquoted for storage. Plasma RBP4 levels will be measured with commercially available ELISA assays.
(Aim 2) Concentration of circulating misfolded TTR oligomers | At baseline for all three cohorts
  Venous blood will be collected by phlebotomy at enrollment for all participants. Circulating misfolded TTR oligomers will be measured with peptide-based probes that selectively label these species in plasma.
(Aim 2) TTR kinetic stability | At baseline for all three cohorts
  Venous blood will be collected by phlebotomy at enrollment for all participants. TTR kinetic stability will be measured by using Western Blot techniques.

OTHER OUTCOMES:
(Sub-aim 2) Associations between each biomarker from Aim 2 and CMRI measurements from Aim 1 and Sub-aim 1 | At baseline for all 3 cohorts and Visit 2 for V122I TTR carriers and age-, sex-, and race-matched controls
  To achieve this, we will employ multivariable generalized linear mixed models to determine the independent association between these biomarkers and CMRI measurements in V122I TTR carriers without HF. Additionally, after determining the univariable association between each biomarker and outcome from Aim 1 and Sub-aim 1, we will employ a backwards selection algorithm from a list of confounders (eGFR, sex, age, hypertension, and BMI) and each biomarker to determine the biomarker(s) most closely associated with subclinical hATTR-CA.

CONTACTS AND LOCATIONS:
Overall Officials: Justin L Grodin, MD MPH, Principal Investigator — UT Southwestern
Locations (3):
- United States (3):
  - Columbia University Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided